CLINICAL TRIAL: NCT04637217
Title: Retinal Neurodegenerative and Vascular Changes in Diabetic Patients: an OCT-based Comparative Study
Brief Title: Retinal Neurodegenerative and Vascular Changes in Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Ioana Damian, Assistant Professor, Iuliu Hatieganu University of Medicine and Pharmacy
Other Study IDs: U1111-1249-7228
Record Dates: First submitted 2020-11-12; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Diabetic Retinopathy; Neurodegeneration
Keywords: optical coherence tomography; choroid; outer retina
MeSH Terms: conditions — Diabetic Retinopathy; Nerve Degeneration | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control
  Interventions: Diagnostic Test: Optical Coherence Tomography
- Diabetes mellitus without Diabetic Retinopathy
  Interventions: Diagnostic Test: Optical Coherence Tomography
- Diabetes mellitus with Diabetic Retinopathy
  Interventions: Diagnostic Test: Optical Coherence Tomography

INTERVENTIONS:
Diagnostic Test: Optical Coherence Tomography — Spectral Domain Optical Coherence Tomography(SD-OCT) examination will be performed for every patient: posterior pole scan, EDI-OCT(enhanced depth imaging-OCT) and peripapillary RNFL(retinal nerve fiber layer)

SUMMARY:
Using Optical Coherence Tomography and ImageJ software the investigators will analyze retinal and choroidal vascular changes and their impact on retinal layers among patients with diabetes without retinopathy and patients with diabetes and retinopathy.

DETAILED DESCRIPTION:
Relieving the burden of diabetic retinopathy treatment require a prompt and non-invasive assessment of diabetic patients before the occurence of diabetic retinopathy. Since OCT is capable of imaging retina with such a high precision, retinal changes occuring before any clinical signs of retinopathy, such as microaneurysm or haemorrhages, can now be assessed. In the present study the investigators are analyzing the connection between retinal arteries and veins regarding lumen diameter, vessel wall thickness and their correlation with retinal nerve fiber layer and ganglion cell layer thickness. Moreover, using binarization of the choroid the investigators will assess its relationship with outer retina layers, such as retinal pigment epithelium and photoreceptors.

ELIGIBILITY:
Inclusion Criteria:

* history of type 1DM for more than 1 year
* history of type 2 DM for more than 3 months
* diagnosis of no DR or mild Non-proliferative diabetic retinopathy(NPDR)

Exclusion Criteria:

* DR with more than NPDR ,
* Diabetic macular oedema,
* media opacities such as corneal or lens opacities that could preclude appropriate OCT imaging,
* presence of other retinal diseases such as Age-related macular degeneration, Vitreo-macular traction, Macular hole, Epiretinal membrane, Retinal vein occlusion, Macular scars,
* Glaucoma, Optic neuropathies or Neurodegenerative diseases,
* history of ocular trauma,
* Refractive errors of more than ±6 diopters (spherical equivalent),
* previous ocular surgery, focal laser, panretinal photocoagulation or anti-VEGF intravitreal injection

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All participants were recruited between July 2018 and July 2019 at Department of Ophthalmology, Emergency County Hospital Cluj, Romania. Healthy subjects were recruited from patients scheduled for routine ocular examination at Department of Ophthalmology, Emergency County Hospital Cluj, Romania
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Correlation between choroid and outer retina using SD-OCT- based binarization technique | 2018-2019
  starting from EDI-OCT scans the investigators will analyze choroidal parameters such as Luminal area, Stromal area, Total choroidal area, Chorodial vascularity index and correlate them with retinal pigment epithelium (RPE),outer nuclear layer(ONL) and photoreceptors' thickness (PR)
Correlation between neurodegeneration and retinal vessels characteristics | 2018-2019
  using full width at half maximum method, the investigators will measure peripapillary arteries and veins' diameters, their wall thickness and correlate them with RNFL and ganglion cell layer(GCL) thickness

SECONDARY OUTCOMES:
Correlation between choroidal parameters and their influence on Best corrected visual acuity(BCVA) | 2018-2019
  The investigators will analyze if changes in the choroid will influence patients' visual acuity. For statistical reasons, visual acuity will be converted to logMAR(logarithm of the minimum angle of resolution)
Correlation between renal function and choroidal parameters | 2018-2019
  Using estimated glomerular filtration rate(eGFR-mL/min/1.73 m2) the investigators will analyze if a decreased eGFR will produce changes in choroidal architecture
Correlation between sistemic factors and choroidal parameters | 2018-2019
  The investigators will document if the presence of High Blood pressure(yes/no) and current smoking(yes/no) influences choroidal thickness or CVI.
Correlation between choroidal parameters and diabetes control | 2018-2019
  Using HbA1c(Glycated haemoglobin) the investigators will analyze the choroidal's behaviour under different HbA1c levels.

CONTACTS AND LOCATIONS:
Overall Officials: Ioana Damian, MD, Principal Investigator — Iuliu Hatieganu University of Medicine and Pharmacy
Locations (1):
- University of Medicine and Pharmacy " Iuliu Hatieganu", Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: After the papers will be published.